CLINICAL TRIAL: NCT03077880
Title: Influence Of Thickness Of the Peri-implant Soft Tissue On Marginal Bone Remodeling Around Bone Level Implant: A Multicenter Observational Clinical Study
Brief Title: Influence of Thickness of the Peri-implant Soft Tissue on Marginal Bone Remodeling
Acronym: STR
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of Piezosurgery Academy, International Piezosurgery Academy
Other Study IDs: STR
Record Dates: First submitted 2017-01-25; First posted 2017-03-13 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Alveolar Bone Loss
Keywords: implant insertion; bone resorption; soft tissue
MeSH Terms: conditions — Alveolar Bone Loss; Bone Resorption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thin soft tissue: full thickness thin mucosal soft tissue at the periodontal probe measured intra-operatory measurement during implant placement
  Interventions: Procedure: intra-operatory measurement during implant placement
- thick soft tissue: full thickness thick mucosal soft tissue at the periodontal probe measured intra-operatory measurement during implant placement
  Interventions: Procedure: intra-operatory measurement during implant placement

INTERVENTIONS:
Procedure: intra-operatory measurement during implant placement — mucoperiosteal flap, soft tissue thickness measurement, implant insertion

SUMMARY:
The aim of this observational study is the evaluation of marginal bone remodeling after surgical implant placement, correlating the gingival thickness with the bone resorption rate.

DETAILED DESCRIPTION:
The present study was designed as a multicenter prospective clinical trial. Five clinical centers will treat patients through the placement of a single dental implant. The fixtures will be prosthetic loaded three months after placement and will be acquired periapical radiographs at each timepoint (base-two months-three-months-6 months-12 months). For every inserted implants the experimental parameters will be collected for the following 2 years.

Surgical procedure. All patients will receive antibiotic prophylaxis with 2 g of amoxicillin one hour before surgery. Crestal incision is performed under local anesthesia with articaine 4% with epinephrine, taking care to preserve the keratinized tissue. With the help of a periosteal elevator, it will be set up carefully buccal flap total thickness, and the vertical thickness of the soft tissue will be measured with a labeled probe every 1.0 mm. If the vertical thickness of the soft tissue will be 2 mm or less, it will be considered thin. If mucosal thickness will be greater than 2 mm, it will be considered thick. After measurement, the lingual flap will be raised to full-thickness, and will be prepared the site for implant placement. The implant site will be at least 1.5 mm from the tooth / teeth adjacent, and must be surrounded by at least 1 mm of bone is buccal to lingual. With a platform switching facility a millimeter will be placed below the level of the bone crest with a one-stage approach as per the manufacturer's recommendations. After insertion, it will be screwed a healing abutment, and the flaps will be sutured without tension with interrupted sutures 4/0. Patients of both groups will be instructed to disinfect the site through a rinse twice a day for a week for 1 minute with 0.12% chlorhexidine digluconate. Patients will be advised to avoid chewing on the operated site and cleaning the healing abutments with an ultra soft toothbrush. After 2 months of healing, it will be evaluated clinical stability and the radiographic appearance of the plants. All plants will be rehabilitated by the prosthetist with single screwed restorations. After the prosthetic treatment, patients will receive oral hygiene instruction and will be monitored through calls to ensure periodontal health (Bleeding on Probing <20% and Plaque Index <25%) throughout the study period.

Radiographic evaluation Intraoral radiographs will be captured in high-resolution mode with a film, customized support from a jig polyvinylsiloxane, using the technique of parallel rays. Intraoral radiographs will be acquired after implant placement (baseline-assessment of inclusion fairness), after 2 months of healing (osseointegration rating), after insertion of the crown (3 months-adaptation assessment of the restoration prosthetic), after 6 months (early loading of evaluation) and after a year of recovery (of the medium-term load rating). The number of intraoral radiographs will be the same which normally is carried out in the course of an implant-prosthetic rehabilitation. The images will be obtained in such a way that the implant-abutment interface is clearly visible. Measurements of bone level will be performed by a blinded central reader using a dedicated program at 20 times magnification. Before the calculation of the crestal bone changes, the RVG images will be calibrated with the implant diameter. bone loss will be calculated by comparing the radiographs at baseline with the radiographs obtained during follow-up visits. The system board and the first contact radiographic bone-implant will be selected as reference points to calculate bone loss. The average of the mesial and distal measurements will be recorded for each implant.

ELIGIBILITY:
Inclusion Criteria:

1. indications for intervention of implant placement in posterior mandible (premolar / molar region) based on a careful diagnosis and treatment plan;
2. presence of a residual osseous crest with a minimum of 7 mm surgical height, and thickness of at least 6 mm at the level of the programmed implant site;
3. the bone crest must be healed (at least 6 months after the loss / extraction of the element corresponding tooth);
4. absence of regenerated bone;
5. plaque index of less than 25% and bleeding index lower than 20%;
6. bucco-lingual width of the attached gingiva ≥ 4 mm;
7. insertion torque plant inserito≥35 N / cm;
8. patient age> 18 years;
9. patients should be able to examine and understand the study protocol;
10. informed consent.

Exclusion Criteria:

1. acute myocardial infarction in the last two months;
2. blood coagulation disorders not compensated;
3. uncontrolled diabetes (HbA1c> 7.5%);
4. radiation therapy of the district head / neck in the last 24 months;
5. immunocompromised patients (HIV infection or chemotherapy) within the last 5 years);
6. present or past treatment with intravenous bisphosphonates;
7. psychological or psychiatric diseases;
8. alcohol or drug abuse;
9. Smoking of local exclusion criteria are the diagnosis of periodontal disease acute or chronic, a previous history of periodontal disease, the presence of regenerated bone, lingual bucco- size of keratinized tissue <4 mm, insertion torque less than 35 N / cm.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients referred to the centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
peri-implant bone resorption | from baseline to twelve months
  radiological assessment of change in the peri-implant bone crest

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr., Principal Investigator — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sicilia A, Quirynen M, Fontolliet A, Francisco H, Friedman A, Linkevicius T, Lutz R, Meijer HJ, Rompen E, Rotundo R, Schwarz F, Simion M, Teughels W, Wennerberg A, Zuhr O. Long-term stability of peri-implant tissues after bone or soft tissue augmentation. Effect of zirconia or titanium abutments on peri-implant soft tissues. Summary and consensus statements. The 4th EAO Consensus Conference 2015. Clin Oral Implants Res. 2015 Sep;26 Suppl 11:148-52. doi: 10.1111/clr.12676. PMID 26385628